CLINICAL TRIAL: NCT01522248
Title: A Pilot Study to Examine the Early Cytokine Responses After Inactivated Influenza Vaccination in Adults 18-50.
Brief Title: Early Immune Responses to Inactivated Influenza Vaccine: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIR 281
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Influenza Virus Vaccine
Keywords: influenza vaccine; cytokines; chemokines; symptoms
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): receives vaccine in morning. Blood drawn at 3, 7, 24, and 48 hours and 14 days after vaccination.
  Interventions: Biological: Trivalent Inactivated Influenza vaccine
- Cohort 2 (Active Comparator): receives vaccine in evening, Blood drawn 16, 40 hours and 14 days after vaccination.
  Interventions: Biological: Trivalent Inactivated Influenza vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza vaccine — 0.5 ml IM once only

SUMMARY:
Some people experience symptoms just after receiving the seasonal inactivated influenza vaccine. The cause of some of these symptoms is likely to be an immune response to the vaccine. The investigators would like to look at the earliest immune responses to the inactivated influenza vaccine. This pilot study will help us to determine at what time points we should look.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-50 years.
2. Good general health as a result of review of medical history and medications.
3. Willingness to participate in the study as evidenced by signing informed consent document.
4. Available for the duration of the trial.

Exclusion Criteria:

1. Known to be pregnant.
2. Medical, behavioral, cognitive or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
3. Severe allergy to eggs or any component of the influenza vaccine
4. Previous receipt of the 2011-2012 season influenza vaccine
5. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the subject unable to comply with the protocol.
6. History of receiving any investigational product within the past 30 days.
7. Participant has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
8. History of a severe allergic reaction or anaphylaxis.
9. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
10. Known immunodeficiency syndrome.
11. Use of chronic (≥14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e. prednisone >10 mg/ day) or immunosuppressive drugs within 30 days of starting this study.
12. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
13. History of a surgical splenectomy.
14. Receipt of blood products within the past 6 months.
15. Refusal to allow storage of samples for future research.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for Immunization Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Talaat KR, Halsey NA, Cox AB, Coles CL, Durbin AP, Ramakrishnan A, Bream JH. Rapid changes in serum cytokines and chemokines in response to inactivated influenza vaccination. Influenza Other Respir Viruses. 2018 Mar;12(2):202-210. doi: 10.1111/irv.12509. Epub 2018 Jan 4. PMID 28991404

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Received vaccine in morning. Blood drawn at 3, 7, 24 and 48 hours and 14 days after vaccination. Trivalent Inactivated Influenza vaccine 0.5ml IM once only
- Cohort 2: Received vaccine in evening. Blood drawn 16 and 40 hours and 14 days after vaccination. Trivalent Inactivated Influenza vaccine 0.5 ml IM once only
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.4) | 35.8 (10.1) | 36.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 3 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Levels of Cytokine Interferon Gamma (IFN-gamma) Responses to Inactivated Influenza Vaccine
Description: This was an exploratory trial to look at the kinetics of early cytokine response to influenza vaccine. Serum collected was assessed for cytokines, and PBMCs may be assessed for innate and adaptive immune responses, as well as for genetic markers associated with immune responses to vaccination. Data for Cohort 1 reported as 0 hours and 24 hours. Data for Cohort 2 reported as 0 hours and 16 hours. Data was combined for the Cohorts and reported as 0 hours (baseline) and 14 days.
Time Frame: 0 hours, 16 hours, 24 hours, 14 days
Population: Data for Cohort 1 reported as 0 hours and 24 hours. Data for Cohort 2 reported as 0 hours and 16 hours. Data was combined for the Cohorts and reported as 0 hours (baseline) and 14 days
Measure: Median (Standard Deviation); unit: pg/mL
Groups:
- Cohort 1: Cytokine Results 0 hours and 24 hours
- Cohort 2: Cytokine results 0hours and 16 hours
- Cohort 1 & 2: Combined Cytokine results 0 hours and 14 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1 & 2
Number analyzed (Participants) | 10 | 10 | 20
pg/mL
  IFN gamma | 1.3 (1.7) | 1.4 (2.2) | 1.3 (1.9)
  IFN-gamma | 6.9 (3.0) | 5.1 (5.0) | 1.2 (0.8)

2. Primary Outcome: Levels of Cytokine Interleukin 8 (IL-8) Cytokine Response to Inactivated Influenza Vaccine
Description: as for outcome 1
Time Frame: 0 hours, 16 hours, 24 hours, 14 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/mL
Groups:
- Cohort 2: Cytokine results 0 hours and 16 hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1 & 2
Number analyzed (Participants) | 10 | 10 | 20
pg/mL
  IL- 8 | 14.7 (7.7) | 11.7 (5.5) | 13.4 (6.9)
  IL-8 | 10.4 (6.1) | 11.9 (4.6) | 10.2 (4.1)

3. Primary Outcome: Levels of Cytokine Interferon Induced Gamma Protein (IP-10) Responses to Inactivated Influenza Vaccine
Description: This was an exploratory trial to look at the kinetics of early (1st 48 hours) cytokine response to influenza vaccine. Serum collected was assessed for cytokines, and PBMCs may be assessed for innate and adaptive immune responses, as well as for genetic markers associated with immune responses to vaccination. Data for Cohort 1 reported as 0 hours and 24 hours. Data for Cohort 2 reported as 0 hours and 16 hours. Data was combined for the Cohorts and reported as 0 hours (baseline) and 14 days.
Time Frame: 0 hours, 16 hours, 24 hours, 14 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: pg/mL
Groups:
- Cohort 1 and 2: Cytokine results 0 hours and 14 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 1 and 2
Number analyzed (Participants) | 10 | 10 | 20
pg/mL
  IP-10 | 115 (74) | 149 (194) | 123 (146)
  IP- 10 | 488 (365) | 292 (309) | 127 (71)

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Cohort 1: Received vaccine in the morning
- Cohort 2: Received vaccine in the evening
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Injection site pain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Diaphoresis (Immune system disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes